CLINICAL TRIAL: NCT05698953
Title: The Effect of Reiki Therapy on Pain, Vital Signs and Quality of Life in Pediatric Oncology Patients
Brief Title: The Effect of Reiki Therapy in Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Duygu Demir, Research Assistant - PhD, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: duygudemir
Record Dates: First submitted 2023-01-02; First posted 2023-01-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Reiki
Keywords: Reiki Touch Therapy; Pediatric Oncology; Pain; Quality of Life; Vital Signs
MeSH Terms: conditions — Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: The study are conducted based on randomized controlled experimental design with double-blind, pre-test-post-test to determine. The research consists of 3 groups. These groups are Reiki group, Placebo group, control group.
Who Masked: Participant
Masking Description: The research consists of 3 groups. These groups are Reiki group, Placebo group, control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki Group (Experimental): Reiki is applied to the Reiki group for 20-30 minutes for three consecutive days.
  Interventions: Other: Reiki
- Placebo Group (Placebo Comparator): Placebo group is applied to the sham Reiki group for 20-30 minutes for three consecutive days Placebo Reiki group is applied to the sham Reiki by an independent nurse during the same application period.
  Interventions: Other: Placebo
- Control Group (No Intervention): No intervention is made in the control group. Standard care was used

INTERVENTIONS:
Other: Reiki — Reiki is applied to the Reiki group for 20-30 minutes for three consecutive days.
  Arms: Reiki Group
Other: Placebo — Placebo group is applied to the sham Reiki group for 20-30 minutes for three consecutive days by an independent nurse during the same application period.
  Other Names: Sham Reiki
  Arms: Placebo Group

SUMMARY:
The study was conducted based on randomized controlled experimental design with double-blind, pre-test-post-test to determine the effect of Reiki applied to pediatric oncology patients aged 5-7 years on pain, vital signs, oxygen saturation (SpO2) and quality of life. While the population of the study consisted of oncology patients aged 5-7 years who were hospitalized in the pediatric oncology services between December 2020 and November 2021, the sample consisted of 66 children diagnosed with leukemia who met the sample selection criteria. The research consists of 3 groups. These groups are Reiki group (n=22), Placebo group (n=22), control group (n=22). The data are collected using Introductory Information Form, Wong-Baker FACES Pain Scale (W-BPS), Vital Signs Follow-up Form, The Pediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module Child and Parent Form. Reiki was applied to the Reiki group for 20-30 minutes for three consecutive days and Placebo was applied to the sham Reiki group by an independent nurse during the same application period. The children in the control group were like the routine of the ward.

DETAILED DESCRIPTION:
The universe of the study consisted of pediatric oncology patients who met the selection criteria in the pediatric oncology services. The study was planned as a randomized controlled experimental design with double-blind, pre-test post-test to determine the effect of Reiki applied to pediatric oncology patients aged 5-7 years on pain, vital signs, oxygen saturation (SpO2) and quality of life. In order for the groups to be distributed homogeneously, the order produced by a computer program (http://www.randomization.com , Balanced permutation) was used. Patients who meet the inclusion criteria and agree to participate in the study assigned to the experimental and control groups according the randomization list. The control variable of the study is demographic characteristics of the children. The dependent variables of the study are pain, vital signs, oxygen saturation parameters and quality of life score.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in the pediatric oncology service at the time of the study
* Being between 5-7 years old
* Body temperature being within normal limits
* To have received at least 1 course of chemotherapy
* Absence of visual, auditory problems or mental retardation at a level that can fill the scales,

Exclusion Criteria:

* To have taken analgesic medication in the last 6 hours,
* Have received any energy and body-mind therapy (yoga, reiki, massage, meditation, healing touch) in the last six months

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the pain score values of the groups | Children's pain levels will be evaluated on the 1st day.
  The Wong-Baker Faces Pain Scale revised (W-BFS) was used to determine the level of pain during the procedure.
  The W-BFS is a scale that is most commonly used in identifying pain in children of the ages 3 to 18. It is reported that the scale is reliable when used with children older than the age of 3 who can verbally express the degree of pain they feel. The scale is made up of faces and numbers. Pain is assessed on a scale of "0" to "10." Pain is described by selecting the facial expression depicting the degree of perceived pain.
Comparison of the pain score values of the groups | Children's pain levels will be evaluated on the 2nd day.
  The Wong-Baker Faces Pain Scale revised (W-BFS) was used to determine the level of pain during the procedure.
  The W-BFS is a scale that is most commonly used in identifying pain in children of the ages 3 to 18. It is reported that the scale is reliable when used with children older than the age of 3 who can verbally express the degree of pain they feel. The scale is made up of faces and numbers. Pain is assessed on a scale of "0" to "10." Pain is described by selecting the facial expression depicting the degree of perceived pain.
Comparison of the pain score values of the groups | Children's pain levels will be evaluated on the 3rd day.
  The Wong-Baker Faces Pain Scale revised (W-BFS) was used to determine the level of pain during the procedure.
  The W-BFS is a scale that is most commonly used in identifying pain in children of the ages 3 to 18. It is reported that the scale is reliable when used with children older than the age of 3 who can verbally express the degree of pain they feel. The scale is made up of faces and numbers. Pain is assessed on a scale of "0" to "10." Pain is described by selecting the facial expression depicting the degree of perceived pain.
Comparison of the heart rate values of the groups | Children's heart rate values will be evaluated on the 1st day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the heart rate values of the children.
Comparison of the heart rate values of the groups | Children's heart rate values will be evaluated on the 2nd day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the heart rate values of the children.
Comparison of the heart rate values of the groups | Children's heart rate values will be evaluated on the 3rd day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the heart rate values of the children.
Comparison of the respiratory rate values of the groups | Children's respiratory rate values will be evaluated on the 1st day.
  The respiratory rate values of the children will be measured by counting for 1 minute.
Comparison of the respiratory rate values of the groups | Children's respiratory rate values will be evaluated on the 2nd day.
  The respiratory rate values of the children will be measured by counting for 1 minute.
Comparison of the respiratory rate values of the groups | Children's respiratory rate values will be evaluated on the 3rd day.
  The respiratory rate values of the children will be measured by counting for 1 minute.
Comparison of the body temperature values of the groups | Children's body temperature values will be evaluated on the 1st day.
  "Cem brand" infrared thermometer device was used to measure body temperature of the children.
Comparison of the body temperature values of the groups | Children's body temperature values will be evaluated on the 2nd day.
  "Cem brand" infrared thermometer device was used to measure body temperature of the children.
Comparison of the body temperature values of the groups | Children's body temperature values will be evaluated on the 3rd day.
  "Cem brand" infrared thermometer device was used to measure body temperature of the children.
Comparison of the oxygen saturation values of the groups | Children's oxygen saturation values will be evaluated on the 1st day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the oxygen saturation values of the children.
Comparison of the oxygen saturation values of the groups | Children's oxygen saturation values will be evaluated on the 2nd day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the oxygen saturation values of the children.
Comparison of the oxygen saturation values of the groups | Children's oxygen saturation values will be evaluated on the 3rd day.
  Finger type portable "Creative PC 60" pulse oximeter device was used to measure the oxygen saturation values of the children.
Comparison of Groups' Quality of Life Scale (PedsQL 3.0 Cancer Module) Scores | Measurements will be made before on the 1st and after 3rd days the intervention.
  The Child and Parent Reports of the PedsQL 3.0 Cancer Module for Young Children (ages 5-7), are composed of 26 items comprising 8 dimensions. Scores are transformed on a scale from 0 to 100. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Higher scores indicate lower problems.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Demir, PhD, Study Chair — Istanbul University - Cerrahpasa; Birsen Mutlu, Assoc. Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- University of Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miles P, True G. Reiki--review of a biofield therapy history, theory, practice, and research. Altern Ther Health Med. 2003 Mar-Apr;9(2):62-72. PMID 12652885
- [Background] Natale GW. Reconnecting to nursing through Reiki. Creat Nurs. 2010;16(4):171-6. doi: 10.1891/1078-4535.16.4.171. PMID 21140870
- [Background] Vitale A. An integrative review of Reiki touch therapy research. Holist Nurs Pract. 2007 Jul-Aug;21(4):167-79; quiz 180-1. doi: 10.1097/01.HNP.0000280927.83506.f6. PMID 17627194
- [Result] Thrane SE, Grossoehme DH, Tan A, Shaner V, Friebert S. Feasibility and Acceptability of a Reiki Intervention With Very Young Children Receiving Palliative Care. Nurs Res. 2021 Nov-Dec 01;70(6):469-474. doi: 10.1097/NNR.0000000000000540. PMID 34262006
- [Result] Thrane SE, Maurer SH, Danford CA. Feasibility and Acceptability of Reiki Therapy for Children Receiving Palliative Care in the Home. J Hosp Palliat Nurs. 2021 Feb 1;23(1):52-58. doi: 10.1097/NJH.0000000000000714. PMID 33252426
- [Result] Thrane SE, Williams E, Grossoehme DH, Friebert S. Reiki Therapy for Very Young Hospitalized Children Receiving Palliative Care. J Pediatr Hematol Oncol Nurs. 2022 Jan-Feb;39(1):15-29. doi: 10.1177/27527530211059435. PMID 35722865
- [Result] Charkhandeh M, Talib MA, Hunt CJ. The clinical effectiveness of cognitive behavior therapy and an alternative medicine approach in reducing symptoms of depression in adolescents. Psychiatry Res. 2016 May 30;239:325-30. doi: 10.1016/j.psychres.2016.03.044. Epub 2016 Mar 30. PMID 27058159
- [Result] Radziewicz RM, Wright-Esber S, Zupancic J, Gargiulo D, Woodall P. Safety of Reiki Therapy for Newborns at Risk for Neonatal Abstinence Syndrome. Holist Nurs Pract. 2018 Mar/Apr;32(2):63-70. doi: 10.1097/HNP.0000000000000251. PMID 29315084
- [Result] Zucchetti G, Candela F, Bottigelli C, Campione G, Parrinello A, Piu P, Vassallo E, Fagioli F. The Power of Reiki: Feasibility and Efficacy of Reducing Pain in Children With Cancer Undergoing Hematopoietic Stem Cell Transplantation. J Pediatr Oncol Nurs. 2019 Sep/Oct;36(5):361-368. doi: 10.1177/1043454219845879. Epub 2019 May 3. PMID 31046557
- [Result] Kocoglu F, Zincir H. The Effect of Reiki on Pain, Fatigue, and Quality of Life in Adolescents With Dysmenorrhea. Holist Nurs Pract. 2021 Nov-Dec 01;35(6):306-314. doi: 10.1097/HNP.0000000000000477. PMID 34647912
- [Result] Vitale AT, O'Connor PC. The effect of Reiki on pain and anxiety in women with abdominal hysterectomies: a quasi-experimental pilot study. Holist Nurs Pract. 2006 Nov-Dec;20(6):263-72; quiz 273-4. PMID 17099413
- [Result] Whelan KM, Wishnia GS. Reiki therapy: the benefits to a nurse/Reiki practitioner. Holist Nurs Pract. 2003 Jul-Aug;17(4):209-17. doi: 10.1097/00004650-200307000-00008. PMID 12889549
- See also: The National Center of Complementary and Alternative Medicine (NCCAM) — http://www.nccih.nih.gov/health/reiki